CLINICAL TRIAL: NCT03077139
Title: Cardiac Resynchronization Therapy in Pulmonary Hypertension
Acronym: CRT in PH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Daniel P Morin, MD MPH FHRS (Other)
Responsible Party: Sponsor-Investigator, Dr. Daniel P Morin, MD MPH FHRS, Cardiac Electrophysiologist, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT in PH
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arms (Experimental): Pacing wires used to stimulate ventricles in a synchronous matter
  Interventions: Device: Cardiac Resynchronization Therapy (CRT)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (CRT) — A CRT device sends small electrical impulses to both lower chambers of the heart to help them beat together in a more synchronized pattern.

SUMMARY:
This study is being conducted to determine whether patients with advanced pulmonary hypertension when treated with cardiac resynchronization therapy improve hemodynamically and/or receive clinical benefit.

DETAILED DESCRIPTION:
This study aims to determine whether stimulating earlier activation of the failing right ventricle in pulmonary hypertension reduces the effects of interventricular dependence in human subjects, thereby improving overall cardiac function and symptoms in patients with pulmonary hypertension and right ventricle failure with NYHA Class 3-4 symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension, defined as pulmonary artery systolic pressure greater than 40 mm Hg by transthoracic echocardiogram or right heart catheterization
* LVEF ≥ 50%
* Baseline 6MWT distant <400 meters
* Baseline NYHA Functional class ≥ III

Exclusion Criteria:

* LVEF < 50%
* 6MWT duration > 400 meters
* NYHA Functional class < III
* Left bundle branch block
* Non-sinus rhythm
* Severe aortic stenosis (Aortic valve area < 1 cm2)
* Severe mitral regurgitation
* Acute cardiac failure
* Dependency on intravenous inotropies
* Severe obstructive pulmonary disease
* Hypertrophic obstructive cardiomyopathy
* Amyloidosis
* Dependence on pacing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
15% increase in cardiac output at the optimal VV interval over baseline cardiac output | the procedure
  Primary Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morin, MD, Principal Investigator — Cardiac Electrophysiologist
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided